CLINICAL TRIAL: NCT02740764
Title: Optimization of Drug Prescribing in an Elderly Population of Geriatric Consultations and Living at Home
Brief Title: Optimization of Drug Prescribing in an Elderly Population of Geriatric Consultations
Acronym: OPTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL15-0104
Record Dates: First submitted 2016-04-06; First posted 2016-04-15 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Functional Autonomy Level
Keywords: Functional autonomy level; Lawton Instrumental Activities of Daily Living; Cognitive disorders; Potentially inappropriate medication; elderly; Optimization of drug prescribing
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimization of drug prescribing (Experimental): The group with optimization program will have: (i) a medical history of the drug prescribing; (ii) analysis and pharmaceutical recommendations and (iii) preparation of a management plan. Notices will be sent only to referring physicians in this experimental group.
  Interventions: Other: Optimization of drug prescribing
- No intervention (No Intervention): This group will receive the current management of patients in geriatric or memory consultation, during which the intervention of a clinician pharmacist is not provided. There will be a history of the drugs prescribing leading to pharmaceutical recommendations by the pharmacist-clinician, accepted by the specialist physicians in charge of the patient at the hospital, but the recommendations will not be transmitted to the referring physicians of patients.

INTERVENTIONS:
Other: Optimization of drug prescribing — The patients included in this group will have the intervention. The optimization of drug prescribing consists to a history of the drugs prescribing leading to pharmaceutical recommendations by the pharmacist-clinician, accepted by the specialist physicians in charge of the patient at the hospital and sent to the referring physicians of patients, who can accept or not the recommendations.
  Arms: Optimization of drug prescribing

SUMMARY:
Aging is often associated with multiple chronic conditions conducting increased consumption of drugs. Drug therapy is necessary for the treatment of many diseases. However, misuse of drugs, particularly linked to the potentially inappropriate prescribing and polypharmacy, increases the iatrogenic risks and can lead to adverse events such as falls, cognitive decline, increased use to the health system: hospital admissions, emergency room visits, and institutionalization. These problems are common since about 20% of emergency room use in elderly patients due to an adverse event related to drugs. Nearly 28% of adverse events related to drug prescriptions could be avoided.

Interventions to optimize drug therapy showed a reduction in the number of potentially inappropriate medications, but their impact on health, has rarely been evaluated. If an association with death has been established, the link with the loss of functional autonomy, which leads to reduced quality of life and significant cost of care, has not been investigated. The evolution towards functional disabilities, frequent with aging has many causes, among which some could be prevented. The optimization of drug prescriptions could thereby delay or prevent the loss of functional autonomy by reducing the risk of adverse events, such as falls or cognitive decline and improving the management of chronic diseases. Our hypothesis is that an optimization program of the drug prescribing may slow progression to functional dependence. To assess the effect of the optimization program of drug prescribing on the level of functional autonomy, a multicenter Randomized Controlled Trial will be conducted in geriatric and memory consultations.

Expected results The implementation of the "OPTIM" program should enable optimization of drug prescribing in elderly patients and therefore slow or prevent progression to addiction. It should also help to develop and strengthen collaboration and communication between the team of geriatric consultation, the clinician pharmacist and referring physicians in town (private practice). In addition, pharmaceutical notice sent to referring physicians should help raise awareness of the prescription of drugs in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and over;
* Patients received for the first time in a geriatric or memory consultation of a study recruiting centers;
* Patients living at home;
* Patients with the ability to express themselves orally or in writing in French sufficiently to carry out clinical assessments;
* Patients who led the last drugs prescription from his referring physician, at the geriatric/memory consultation (in current practice, patients should take the last prescription established by the referring physician);
* Patients accompanied by a caregiver.

Exclusion Criteria:

* Patients with no discernment;
* Patient put under legal protection;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 302 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
The evolution of the level of functional autonomy of the patients assessed using the scale IADL of Lawton | At inclusion
  The primary outcome will be calculated using the 4 successive evaluations of IADL scale.
  The IADL scale assesses the level of functional autonomy of a patient through the assessment of instrumental activities of daily living: ability to use the telephone, transportation, shopping, managing medications, manage a budget, prepare meals, maintain the house and do the laundry. The rating scale provides a score from 0 to 8. A higher score indicates a higher level of dependency, while a lower score reflects a lower level of dependence. The IADL scale consists of 8 questions.
The evolution of the level of functional autonomy of the patients assessed using the scale IADL of Lawton | At 1 month
  The primary outcome will be calculated using the 4 successive evaluations of IADL scale.
The evolution of the level of functional autonomy of the patients assessed using the scale IADL of Lawton | At 6 months
  The primary outcome will be calculated using the 4 successive evaluations of IADL scale.
The evolution of the level of functional autonomy of the patients assessed using the scale IADL of Lawton | At 18 months
  The primary outcome will be calculated using the 4 successive evaluations of IADL scale.
The evolution of the level of functional autonomy of the patients assessed using the scale DAD-6. | At inclusion
  The primary outcome will be calculated using the 4 successive evaluations of DAD-6 scale.
  The scale DAD-6 assesses the patient's activities in his daily life. It includes six questions assessing the degree of autonomy for the following activities: Food, use the telephone or the computer, moving outside, finance and correspondence, medications, leisure and home maintenance. The score ranges from 0 to 18 points, the higher the score, the more the patient is autonomous.
The evolution of the level of functional autonomy of the patients assessed using the scale DAD-6. | At 1 month
  The primary outcome will be calculated using the 4 successive evaluations of DAD-6 scale.
  The scale DAD-6 assesses the patient's activities in his daily life. It includes six questions assessing the degree of autonomy for the following activities: Food, use the telephone or the computer, moving outside, finance and correspondence, medications, leisure and home maintenance. The score ranges from 0 to 18 points, the higher the score, the more the patient is autonomous.
The evolution of the level of functional autonomy of the patients assessed using the scale DAD-6. | At 6 months
  The primary outcome will be calculated using the 4 successive evaluations of DAD-6 scale.
  The scale DAD-6 assesses the patient's activities in his daily life. It includes six questions assessing the degree of autonomy for the following activities: Food, use the telephone or the computer, moving outside, finance and correspondence, medications, leisure and home maintenance. The score ranges from 0 to 18 points, the higher the score, the more the patient is autonomous.
The evolution of the level of functional autonomy of the patients assessed using the scale DAD-6. | At 18 months
  The primary outcome will be calculated using the 4 successive evaluations of DAD-6 scale.
  The scale DAD-6 assesses the patient's activities in his daily life. It includes six questions assessing the degree of autonomy for the following activities: Food, use the telephone or the computer, moving outside, finance and correspondence, medications, leisure and home maintenance. The score ranges from 0 to 18 points, the higher the score, the more the patient is autonomous.

SECONDARY OUTCOMES:
Number of Hospitalizations | Baseline, 1 month, 6 months and 18 months
  the occurrence of hospitalizations within 18 months after baseline
Number of days before hospitalizations | Baseline, 1 month, 6 months and 18 months
  delay between baseline and the hospitalization
Occurrence of recourse to emergency service | Baseline, 1 month, 6 months and 18 months
  occurrence of recourse to emergency service within 18 months after baseline
Number of days before the recourse to emergency service | Baseline, 1 month, 6 months and 18 months
  delay between baseline and the recourse to emergency service
The occurrence of admission in institution | Baseline, 1 month, 6 months and 18 months
  the occurrence of admission in institution within 18 months after baseline
Number of days before admission in institution | Baseline, 1 month, 6 months and 18 months
  delay between baseline and the admission in institution
Death | Baseline, 1 month, 6 months and 18 months
  the occurrence of death within 18 months after baseline
Number of days before death | Baseline, 1 month, 6 months and 18 months
  delay between baseline and death
Falls | Baseline, 1 month, 6 months and 18 months
  the occurrence of falls within 18 months after baseline
Number of days before falls | Baseline, 1 month, 6 months and 18 months
  the delay between baseline and falls
Cognitive functions | Baseline, 6 months and 18 months
  The cognitive function is measured by the Mini Mental State Examination (MMSE) at every visit, as part of the routine care pathway of the patient. Successive scores will be used to measure the evolution of MMSE.
Quality of life 1 | Baseline, 6 months and 18 months
  Quality of life measured by questionnaire QoL-AD
Quality of life 2 | Baseline, 6 months and 18 months
  Quality of life measured by questionnaire EUROQOL 5D
depression disorders | Baseline, 6 months and 18 months
  depression measured with the mini-GDS scale
Anxiety disorders | Baseline, 6 months and 18 months
  Anxiety disorders will be measured with the Hamilton scale
Compliance of patients with treatment | Baseline, 6 months and 18 months
  compliance is measured with the questionnaire Girerd
Pain | Baseline, 6 months and 18 months
  Pain is measured with an ordinal scale from 0 to 10
Proportion of potential inappropriate medication | Baseline, 1 month, 6 months and 18 months
  The proportion of potential inappropriate medication will be measured on the drug prescribing of the patients issued from the referring physician
Problems associated with drug therapy | Baseline, 1 month, 6 months and 18 months
  The proportion of problems associated with drug therapy will be measured on the drugs prescribing of the patients issued from the referring physician
acceptance rate by the referring physicians of pharmaceutical recommendation | Baseline, 1 month, 6 months and 18 months
  The acceptance rate of the pharmaceutical review will be evaluated in 2 complementary ways:
  * By comparing patients' prescriptions issued by the referring physician before and after the pharmaceutical review.
  * By interviewing the referring physician

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital gériatrique du Mont d'Or, Albigny-sur-Saône
  - Hôpital des Charpennes, Lyon

REFERENCES:
- [Derived] Dauphinot V, Jean-Bart E, Krolak-Salmon P, Mouchoux C. A multi-center, randomized, controlled trial to assess the efficacy of optimization of drug prescribing in an elderly population, at 18 months of follow-up, in the evolution of functional autonomy: the OPTIM study protocol. BMC Geriatr. 2017 Aug 30;17(1):195. doi: 10.1186/s12877-017-0600-7. PMID 28854884